CLINICAL TRIAL: NCT02732834
Title: Clinician-Patient Communication in Lung Cancer Care
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hamad Medical Corporation (Industry); University of Arizona (Other); Weill Medical College of Cornell University (Other); University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 16-001
Record Dates: First submitted 2016-03-14; First posted 2016-04-11 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer
Keywords: Clinician-Patient Communication; 16-001
MeSH Terms: conditions — Lung Neoplasms | interventions — Surveys and Questionnaires; Patient Selection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Part 1: Lung patients: Following informed consent, the patient will complete the patient questionnaire, either electronically, by phone, or on paper. Patients who prefer to complete the survey electronically will be emailed a link to access to a secure electronic (web-based) version of the study assessment which they will have access to from any computer. We will include an introductory email with the survey link. Will audio-record actual patient-physician clinical consultations with lung cancer patients at Memorial Sloan Kettering (MSK). Completing the survey will take about 15 minutes. Answer a few open-ended questions about the consultation with the doctor. We will audio record your answers to these questions. This will take about 15 minutes.
  Interventions: Behavioral: Questionnaire; Behavioral: Patient Interview; Behavioral: Audio recordings of clinical consultations
- Part 1: Thoracic physicians and clinicians: Will have 5 visits/consultations with their patients audio recorded.
  Interventions: Behavioral: Audio recordings of clinical consultations
- Part 2: Lung patients: Following informed consent, the patient will complete the patient questionnaire, either electronically, by phone, or on paper. Patients who prefer to complete the survey electronically will be emailed a link to access to a secure electronic (web-based) version of the study assessment which they will have access to from any computer. Completing the survey will take about 15 minutes.
  Interventions: Behavioral: Questionnaire
- Part 2: Thoracic and pulmonary clinicians: Following informed consent, clinicians will be scheduled to participate in a 2 hour training on empathic communication with lung cancer patients. Surveys will be collected from 6 patients (3 pre-training, 3 post-training). Clinicians will complete one standardized patient assessment before training (pre-SPA) and one assessment after training (post-SPA). These are 12-minute video-recorded clinic consultations with standardized patients (trained actors).
  Interventions: Behavioral: 2-hour empathic communication skills training; Behavioral: Standardized Patient Assessments; Behavioral: Training evaluation; Behavioral: Patient recruitment

INTERVENTIONS:
Behavioral: Questionnaire — patients will fill out a questionnaire about their perceived stigma, satisfaction with communication, and psychological distress.
  Groups: Part 1: Lung patients
Behavioral: Patient Interview — Then they will participate in a brief in-person interview about their perceived stigma during the clinical consultation
  Groups: Part 1: Lung patients
Behavioral: Audio recordings of clinical consultations
  Groups: Part 1: Lung patients; Part 1: Thoracic physicians and clinicians
Behavioral: Questionnaire — Patients will fill out a questionnaire about their perceived stigma and satisfaction with their clinician's communication.
  Groups: Part 2: Lung patients
Behavioral: 2-hour empathic communication skills training — 2-hour empathic communication skills training
  Groups: Part 2: Thoracic and pulmonary clinicians
Behavioral: Standardized Patient Assessments — pre-training SPA, post-training SPA
  Groups: Part 2: Thoracic and pulmonary clinicians
Behavioral: Training evaluation — Clinicians will complete an evaluation assessing the empathic communication training module.
  Groups: Part 2: Thoracic and pulmonary clinicians
Behavioral: Patient recruitment — 6 of the clinician's patients (3 pre-training, 3 post-training) will be recruited to complete brief surveys assessing clinician communication
  Groups: Part 2: Thoracic and pulmonary clinicians

SUMMARY:
The purpose of this study is to better understand communication between patients with lung cancer and their clinicians. The investigators are also interested in patient's perceptions of the quality of communication with his/her clinician and how these perceptions may impact patient outcomes. The clinician participating in this study and has given us permission to approach his/her eligible patients for study participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed lung cancer diagnosis or mass suspicious of lung cancer as per clinician report and/or EMR
* Lung cancer diagnosis or suspicious mass as per clinician report/EMR within 0-6 months of consent or within no more than three visits to participating clinician
* Participating clinician approves his/her patient's participation in this study per clinician report.
* Former (at least 100 cigarettes in lifetime and quit more than 30 days prior to enrollment) or current smoker (lifetime smoker who reports cigarette smoking within the past 30 days) as per self report or EMR;
* English fluency (determined through EMR or clinician report), as we do not have the resources to translate the consultations from other languages or the surveys to other languages;
* Patients must be 18 years old or older

Clinician Inclusion Criteria:

* An MSK attending physician (radiologists, medical oncologists, and surgeons), Nurse Practitioner (NP), Physician Assistant (PA), Fellow, Resident or Clinical Nurse Specialist (CNS) or Clinical Nurse (RN) who is a member of the Thoracic Disease Management Team or Pulmonary Service currently treating thoracic patients at MSK as per self report
* Clinical has individual clinic consultations to discuss adult health assessment and/or smoking history with the target patient population: English-speaking, at least 18 years of age, has a suspicious lung mass or confirmed diagnosis, is a former/current smoker, has had no more than 3 visits with clinician or had diagnosis in past 6 months as per self-report.

Exclusion Criteria:

Clinician Exclusion Criteria

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MSK thoracic clinic, pulmonary clinic
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Part 1: Systematic coding of clinical encounters and the perceived stigma within the clinical consultation | 1 year
  interview along with patient-reported data from the post-consultation questionnaire will be used.
Part 1: All variables (stigma, satisfaction with communication, psychological distress) | 1 year
  will be measured via post-consultation questionnaires
Part 2: We will pilot test the effectiveness of the empathic communication skills training module | 1 year
  for clinicians: physicians, nurse practitioners, physician assistants, fellows, residents, clinical nurses, and clinical nurse specialists by using the communication skills training module

SECONDARY OUTCOMES:
# of patients referred to MSK's Tobacco Treatment Program (TTP) | 1 year
  will be determined via review of the medical record and/or Tobacco Treatment Program database

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and follow-up only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent and follow-up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and follow-up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and follow-up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and follow-up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT02732834/ICF_000.pdf